CLINICAL TRIAL: NCT00141921
Title: An Open-Label Extension Study to Evaluate the Safety of Etanercept in Pediatric Subjects With Plaque Psoriasis
Brief Title: Pediatric Open-Label Extension Study of Etanercept in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050111
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Pediatric Plaque Psoriasis
Keywords: Immunex; Amgen; Pediatric,; plaque psoriasis; clinical trial
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept (Experimental): Participants received etanercept 0.8 mg/kg (up to a maximum dose of 50 mg) once weekly by subcutaneous injection for up to 264 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Open-label at a dose of 0.8 mg/kg (up to an intended dose of 50 mg) given once weekly by subcutaneous injection
  Other Names: Enbrel®

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of etanercept in pediatric patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
This study was a multicenter, open-label extension study for pediatric patients who participated in Study 20030211 (NCT00078819).

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on previous Amgen study 20030211 (NCT00078819)

Exclusion Criteria:

* Serious or clinically significant adverse event on Amgen study 20030211 related to etanercept

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2005-08-11 (Actual); Primary Completion 2011-12-19 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Paller AS, Siegfried EC, Eichenfield LF, Pariser D, Langley RG, Creamer K, Kricorian G. Long-term etanercept in pediatric patients with plaque psoriasis. J Am Acad Dermatol. 2010 Nov;63(5):762-8. doi: 10.1016/j.jaad.2010.04.004. Epub 2010 Jun 3. PMID 20605256
- [Background] Paller AS, Siegfried EC, Pariser DM, Rice KC, Trivedi M, Iles J, Collier DH, Kricorian G, Langley RG. Long-term safety and efficacy of etanercept in children and adolescents with plaque psoriasis. J Am Acad Dermatol. 2016 Feb;74(2):280-7.e1-3. doi: 10.1016/j.jaad.2015.09.056. PMID 26775775
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed to evaluate the long-term safety and efficacy of etanercept in pediatric patients with moderate to severe plaque psoriasis who participated in Study 20030211 (NCT00078819).
  The study was conducted at 38 sites in the United States and Canada.
Pre-assignment Details: Results reported below are from the main analysis performed at year 5 (264 weeks).
Period: Overall Study
Arm/Group | Etanercept
Started | 182
Received Treatment | 181
Completed | 41
Not Completed | 141
Not completed — Remain on Study | 28
Not completed — Withdrawal by Subject | 42
Not completed — Lost to Follow-up | 19
Not completed — Noncompliance | 17
Not completed — Disease Progression | 7
Not completed — Protocol Deviation | 7
Not completed — Adverse Event | 5
Not completed — Administrative Decision | 2
Not completed — Pregnancy | 4
Not completed — Ineligibility Determined | 2
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 92
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 138
  Black or African American | 10
  Hispanic or Latino | 17
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 1
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse events is any AE that
  * is fatal
  * is life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * other significant medical hazard. The severity assessment for adverse events and infections (except injection site reactions) was done using the Common Toxicity Criteria (CTC) Version 2.0, where Grade 3 indicates a severe toxicity (incapacitating with inability to work or do usual activity).
  An infectious event is an event that was considered by the investigator to be an infectious episode. An injection site reaction is a reaction at the site of the subcutaneous injection, commonly characterized, but not limited to symptoms of erythema (redness, usually raised), pruritis (itching), swelling, or pain that is persistent for 4 hours or longer.
Time Frame: 264 Weeks
Population: Participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
participants
  Any adverse event | 161
  Non-infectious adverse events | 149
  Infections | 140
  Grade 3 non-infectious adverse events | 14
  Grade 3 infections | 5
  Serious non-infectious adverse events | 5
  Serious infections | 2
  Non-infectious AEs leading to study withdrawal | 5
  Infections leading to withdrawal from study | 1
  Injection site reactions | 16
  Deaths | 0

2. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: An injection site reaction is a reaction at the site of the subcutaneous injection, commonly characterized, but not limited to symptoms of erythema (redness, usually raised), pruritis (itching), swelling, or pain that is persistent for 4 hours or longer.
Time Frame: 264 weeks
Population: Participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
participants
  Any injection site reaction | 16
  Injection site erythema | 6
  Injection site reaction | 4
  Injection site pruritus | 3
  Injection site haematoma | 2
  Injection site swelling | 2
  Injection site discolouration | 1
  Injection site irritation | 1
  Injection site pain | 1

3. Secondary Outcome: Exposure-adjusted Adverse Event Rates
Description: The exposure adjusted event rate for a given event in a given time period is defined as the number of events reported in the given time period divided by total patient-years on investigational product during the period.
  Exposure-adjusted event rate per 100 patient years = total number of events / patient years * 100.
  Multiple occurrences of the same event for a participant were counted as multiple events.
Time Frame: 264 weeks
Population: Participants who received at least one dose of investigational product.
Measure: Number; unit: events per 100 patient years
Arm/Group | Etanercept
Number analyzed (Participants) | 181
events per 100 patient years
  All adverse events | 215.8
  Non-infectious Adverse Events | 115.9
  Infections | 97.3
  Injection Site Reactions | 2.6

4. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Time Frame: 264 weeks
Population: Participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
participants | 0

5. Secondary Outcome: Number of Participants With Grade 3 and 4 Laboratory Toxicities
Description: The severity assessment for adverse events and infections (not including injection site reaction) used the Common Toxicity Criteria (CTC) Version 2.0, where Grade 1= Mild - aware of sign or symptom, but easily tolerated; Grade 2= Moderate - discomfort enough to cause interference with usual activity; Grade 3 = Severe - incapacitating with inability to work or do usual activity; Grade 4= Life-threatening - refers to an event in which the patient was, in the view of the investigator, at risk of immediate death at the time of event; Grade 5 = Fatal.
Time Frame: 264 weeks
Population: Participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
participants
  Grade 3 high creatinine | 1
  Grade 3 high hemoglobin | 1
  Grade 3 low hemoglobin | 1
  Grade 3 high alanine aminotransferase | 1
  Grade 3 high white blood cells | 1
  Any grade 4 toxicity | 0

6. Secondary Outcome: Number of Participants Who Developed Anti-etanercept Antibodies
Description: Binding antibodies to etanercept were detected using an anti-etanercept immunoassay. The positive samples in the immunoassay were further analyzed for the presence of neutralizing antibodies using a bioassay.
  Participants who developed anti-etanercept antibodies are those who were antibody positive post-baseline with a negative or no result at baseline.
Time Frame: 264 weeks
Population: Participants who received at least one dose of investigational product and had a post-baseline antibody result.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 169
participants
  Binding antibody positive | 18
  Neutralizing antibody positive | 0

7. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 50 Response (PASI 50)
Description: A PASI 50 response is a 50% or greater improvement (reduction) from baseline in PASI score.
  The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and weeks 12, 48, 96, 144, 192, 240 and 264
Population: Participants who received at least one dose of investigational product and with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
percentage of participants
  Week 12 (N = 181) | 89.5
  Week 48 (N = 168) | 89.3
  Week 96 (N = 138) | 89.1
  Week 144 (N = 114) | 88.6
  Week 192 (n = 92) | 87.0
  Week 240 (N = 74) | 91.9
  Week 264 (N = 66) | 87.9

8. Secondary Outcome: Percentage of Participants With a PASI 75 Response
Description: A PASI 75 response is a 75% or greater improvement (reduction) from baseline in PASI score.
  The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and weeks 12, 48, 96, 144, 192, 240 and 264
Population: Participants who received at least one dose of investigational product with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
percentage of participants
  Week 12 (N = 181) | 67.4
  Week 48 (N = 168) | 67.3
  Week 96 (N = 138) | 60.9
  Week 144 (N = 114) | 62.3
  Week 192 (n = 92) | 69.6
  Week 240 (N = 74) | 64.9
  Week 264 (N = 66) | 63.6

9. Secondary Outcome: Percentage of Participants With a PASI 90 Response
Description: A PASI 90 response is a 90% or greater improvement (reduction) from baseline in PASI score.
  The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and weeks 12, 48, 96, 144, 192, 240 and 264
Population: Participants who received at least one dose of investigational product with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
percentage of participants
  Week 12 (N = 181) | 35.4
  Week 48 (N = 168) | 32.7
  Week 96 (N = 138) | 29.7
  Week 144 (N = 114) | 28.1
  Week 192 (n = 92) | 35.9
  Week 240 (N = 74) | 36.5
  Week 264 (N = 66) | 28.8

10. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in PASI Score
Description: The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 12, 48, 96, 144, 192, 240 and 264
Population: Participants who received at least one dose of investigational product with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 181
percent improvement
  Study 20050111 baseline (N = 179) | 74.429 (22.146)
  Week 12 (N = 181) | 78.286 (21.079)
  Week 48 (N = 168) | 77.546 (20.682)
  Week 96 (N = 138) | 75.355 (24.139)
  Week 144 (N = 114) | 75.052 (23.839)
  Week 192 (n = 92) | 77.815 (23.965)
  Week 240 (N = 74) | 78.924 (23.497)
  Week 264 (N = 66) | 74.605 (29.327)

11. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1)
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). A sPGA response is defined as a sPGA value of clear (score 0) or almost clear (score 1).
Time Frame: Weeks 12, 48, 96, 144, 192, 240 and 264
Population: Participants who received at least one dose of investigational product with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 181
percentage of participants
  Week 12 (N = 181) | 53.6
  Week 48 (N = 168) | 48.8
  Week 96 (N = 139) | 47.5
  Week 144 (N = 114) | 45.6
  Week 192 (n = 92) | 47.8
  Week 240 (N = 74) | 50.0
  Week 264 (N = 66) | 37.9

12. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in Children's Dermatology Life Quality Index (CDLQI) Total Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (Not at all) to 3 (Very much). The total score ranges from 0 to 30, with lower scores indicating better quality of life. If participants were ≥ 13 years old, the text instrument was completed by the participants themselves. Participants ≥ 8 but < 13 years old used the cartoon version of the instrument and participants ≤ 7 years old used the cartoon version of the instrument completed with help from the parents or caregivers.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: Participants who received at least one dose of investigational product with baseline data, and with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 173
percent improvement
  Study 20050111 baseline (N = 164) | 59.492 (73.501)
  Week 24 (N = 155) | 54.978 (69.744)
  Week 48 (N = 148) | 59.229 (65.259)
  Week 72 (N = 136) | 57.549 (79.389)
  Week 96 (N = 127) | 61.084 (66.169)
  Week 120 (N = 105) | 64.059 (75.298)
  Week 144 (N = 103) | 69.732 (42.008)
  Week 168 (N = 93) | 67.531 (42.261)
  Week 192 (N = 81) | 65.622 (53.359)
  Week 216 (N = 70) | 76.121 (43.217)
  Week 240 (N = 64) | 73.631 (54.704)
  Week 264 (N = 56) | 63.291 (63.555)

13. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in CDLQI Symptoms and Feelings Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (not at all) to 3 (Very much). The CDLQI Symptoms and Feelings Score includes 2 questions and ranges from 0 to 6, with lower scores indicating better quality of life.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: Participants who received at least one dose of investigational product with baseline data and with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 173
percent improvement
  Study 20050111 baseline (N = 165) | 54.869 (56.213)
  Week 24 (N = 155) | 55.366 (64.039)
  Week 48 (N = 149) | 53.792 (65.857)
  Week 72 (N = 136) | 51.005 (68.117)
  Week 96 (N = 128) | 55.430 (57.430)
  Week 120 (N = 105) | 53.302 (67.555)
  Week 144 (N = 104) | 56.250 (58.194)
  Week 168 (N = 94) | 58.901 (49.431)
  Week 192 (N = 81) | 55.700 (56.352)
  Week 216 (N = 71) | 71.056 (41.396)
  Week 240 (N = 65) | 67.538 (43.418)
  Week 264 (N = 57) | 56.725 (52.965)

14. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in CDLQI Leisure Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (not at all) to 3 (Very much). The CDLQI Leisure Score includes 3 questions and ranges from 0 to 9, with lower scores indicating better quality of life.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 173
percent improvement
  Study 20050111 baseline (N = 165) | 51.088 (52.612)
  Week 24 (N = 156) | 50.546 (58.606)
  Week 48 (N = 148) | 51.792 (61.204)
  Week 72 (N = 136) | 50.792 (70.769)
  Week 96 (N = 129) | 48.686 (68.482)
  Week 120 (N = 105) | 59.031 (49.472)
  Week 144 (N = 104) | 57.125 (54.284)
  Week 168 (N = 94) | 55.198 (52.141)
  Week 192 (N = 81) | 47.989 (72.947)
  Week 216 (N = 71) | 58.545 (60.440)
  Week 240 (N = 64) | 55.727 (64.420)
  Week 264 (N = 56) | 50.072 (62.049)

15. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in CDLQI School or Holidays Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (not at all) to 3 (Very much). The CDLQI School or Holidays Score includes 1 question (How much did your skin problem effect your school work/holiday plans over the last week?) and ranges from 0 to 3, with lower scores indicating better quality of life.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 173
percent improvement
  Study 20050111 baseline (N = 165) | 31.616 (51.981)
  Week 24 (N = 156) | 32.585 (52.750)
  Week 48 (N = 148) | 36.149 (51.778)
  Week 72 (N = 133) | 29.825 (53.025)
  Week 96 (N = 129) | 29.457 (55.805)
  Week 120 (N = 105) | 32.063 (55.166)
  Week 144 (N = 105) | 33.333 (48.371)
  Week 168 (N = 94) | 32.979 (50.563)
  Week 192 (N = 81) | 31.070 (52.886)
  Week 216 (N = 71) | 35.211 (48.103)
  Week 240 (N = 65) | 26.923 (56.649)
  Week 264 (N = 57) | 27.193 (51.815)

16. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in CDLQI Personal Relationships Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (not at all) to 3 (Very much). The CDLQI Personal Relationships Score includes 2 questions and ranges from 0 to 6, with lower scores indicating better quality of life.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 173
percent improvement
  Study 20050111 baseline (N = 166) | 45.452 (65.038)
  Week 24 (N = 156) | 49.797 (59.328)
  Week 48 (N = 149) | 50.895 (60.179)
  Week 72 (N = 136) | 54.669 (54.519)
  Week 96 (N = 129) | 48.346 (60.414)
  Week 120 (N = 105) | 51.206 (54.435)
  Week 144 (N = 105) | 50.365 (49.636)
  Week 168 (N = 94) | 44.557 (72.287)
  Week 192 (N = 81) | 52.284 (56.125)
  Week 216 (N = 71) | 61.737 (48.255)
  Week 240 (N = 65) | 56.282 (52.042)
  Week 264 (N = 57) | 56.140 (52.481)

17. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in CDLQI Sleep Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (not at all) to 3 (Very much). The CDLQI Sleep Score includes 1 question (How much has your sleep been affected by your skin problems over the last week?) and ranges from 0 to 3, with lower scores indicating better quality of life.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 171
percent improvement
  Study 20050111 baseline (N = 161) | 36.646 (56.851)
  Week 24 (N = 153) | 36.057 (60.349)
  Week 48 (N = 144) | 31.597 (56.329)
  Week 72 (N = 132) | 34.596 (57.390)
  Week 96 (N = 127) | 32.940 (55.216)
  Week 120 (N = 101) | 29.538 (61.503)
  Week 144 (N = 102) | 41.013 (50.229)
  Week 168 (N = 93) | 37.814 (49.888)
  Week 192 (N = 81) | 34.774 (54.658)
  Week 216 (N = 71) | 35.681 (50.811)
  Week 240 (N = 65) | 39.231 (48.808)
  Week 264 (N = 56) | 36.012 (57.890)

18. Secondary Outcome: Percent Improvement From Study 20030211 Baseline in CDLQI Treatment Satisfaction Score
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (not at all) to 3 (Very much). The CDLQI Treatment Satisfaction Score includes 1 question (How much of a problem has the treatment for your skin been over the last week?) and ranges from 0 to 3, with lower scores indicating better quality of life.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 and 264
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Etanercept
Number analyzed (Participants) | 169
percent improvement
  Study 20050111 baseline (N = 161) | 23.085 (64.713)
  Week 24 (N = 152) | 13.268 (74.987)
  Week 48 (N = 144) | 18.634 (67.750)
  Week 72 (N = 134) | 23.383 (73.210)
  Week 96 (N = 128) | 17.969 (72.561)
  Week 120 (N = 105) | 17.778 (65.709)
  Week 144 (N = 104) | 21.795 (62.924)
  Week 168 (N = 93) | 20.430 (73.849)
  Week 192 (N = 81) | 26.955 (68.443)
  Week 216 (N = 71) | 31.455 (59.598)
  Week 240 (N = 65) | 30.513 (57.703)
  Week 264 (N = 56) | 37.500 (64.842)

19. Secondary Outcome: Improvement From Study 20030211 Baseline in Joint Pain
Description: Participants were asked to indicate how much joint pain they had experienced in the last 7 days on a visual analog scale (VAS) from no pain on the left end of the line (score = 0) to severe pain on the right side of the line (score = 10).
  Improvement from baseline = (Baseline Value - Post-baseline Value).
Time Frame: Study 20030211 baseline, Study 20050111 baseline and weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252 and 264
Population: Participants who received at least one dose of investigational product and who completed the joint pain assessment at Study 20030211 baseline, and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 41
units on a scale
  Study 20050111 baseline (N = 31) | 1.5 (2.7)
  Week 12 (N = 29) | 2.3 (2.5)
  Week 24 (N = 22) | 2.4 (3.2)
  Week 36 (N = 22) | 1.5 (3.2)
  Week 48 (N = 24) | 1.5 (3.5)
  Week 60 (N = 14) | 1.3 (3.2)
  Week 72 (N = 16) | 2.1 (3.6)
  Week 84 (N = 14) | 2.9 (3.0)
  Week 96 (N = 16) | 2.0 (2.7)
  Week 108 (N = 14) | 2.4 (3.4)
  Week 120 (N = 12) | 2.4 (2.9)
  Week 132 (N = 15) | 1.9 (3.7)
  Week 144 (N = 12) | 1.8 (4.3)
  Week 156 (N = 12) | 2.5 (3.8)
  Week 168 (N = 10) | 2.2 (4.0)
  Week 180 (N = 11) | 2.7 (3.3)
  Week 192 (N = 11) | 2.5 (4.2)
  Week 204 (N = 11) | 2.8 (3.6)
  Week 216 (N = 9) | 2.9 (3.4)
  Week 228 (N = 10) | 2.8 (3.6)
  Week 240 (N = 9) | 2.7 (3.4)
  Week 252 (N = 8) | 3.9 (3.7)
  Week 264 (N = 8) | 3.9 (3.3)

ADVERSE EVENTS:
Time Frame: 264 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 7/181
Other Adverse Events (participants affected / at risk) | 148/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=181)
Thyroid cyst (Endocrine disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Abortion induced (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=181)
Abdominal pain upper (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 13
Pyrexia (General disorders) | 17
Bronchitis (Infections and infestations) | 18
Ear infection (Infections and infestations) | 12
Gastroenteritis (Infections and infestations) | 14
Gastroenteritis viral (Infections and infestations) | 14
Influenza (Infections and infestations) | 21
Nasopharyngitis (Infections and infestations) | 47
Pharyngitis (Infections and infestations) | 15
Pharyngitis streptococcal (Infections and infestations) | 27
Sinusitis (Infections and infestations) | 24
Upper respiratory tract infection (Infections and infestations) | 68
Urinary tract infection (Infections and infestations) | 12
Viral upper respiratory tract infection (Infections and infestations) | 11
Ligament sprain (Injury, poisoning and procedural complications) | 11
Procedural pain (Injury, poisoning and procedural complications) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24
Headache (Nervous system disorders) | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20
Acne (Skin and subcutaneous tissue disorders) | 33
Dermatitis contact (Skin and subcutaneous tissue disorders) | 11
Psoriasis (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.